CLINICAL TRIAL: NCT06609707
Title: Tuning in to Kids: A Virtually-delivered, Group-based, Psychological Intervention for Parents to Improve Emotional and Behavioral Wellbeing Among Children With Congenital Heart Disease
Brief Title: Tuning in to Kids: An Online, Group Program Tailored for Parents of Children With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Nadine Kasparian, Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0337
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Defects, Congenital; Parenting; Emotion Regulation
Keywords: Congenital Heart Disease; Mental Health; Parenting; Psychological Intervention; Randomized Controlled Trial; Parent Mental Health; Child Mental Health; Emotion Coaching; Parent-Focused Intervention
MeSH Terms: conditions — Heart Defects, Congenital; Emotional Regulation; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Cardiac Care (No Intervention): Participants assigned to the Standard Cardiac Care group will continue to participate in their child's usual cardiac care and can access any supports available to their child and family. Participants in this group will not take part in the Tuning in to Kids program as part of this study; however, once the study has ended, participants will be offered an opportunity to receive Tuning in to Kids, if they would like to.
- Tuning in to Kids (Treatment Arm) (Experimental): Participants will receive Standard Cardiac Care plus the Tuning in to Kids intervention.
  Interventions: Behavioral: Tuning in to Kids

INTERVENTIONS:
Behavioral: Tuning in to Kids — Tuning in to Kids is an evidence-based, emotion-focused, group parenting program designed to teach caregivers skills in recognizing, understanding, and managing their own and their children's emotions. The program includes six 90-minute, weekly, online group sessions and two optional 'booster' sessions to consolidate skills. Parents are taught five steps of emotion coaching and participate in exercises sequentially targeting each step. Intervention components include psychoeducation, emotion coaching demonstrations, role plays, group discussion, written resources, and home practice exercises. The program teaches parents skills in emotion coaching as a way of responding to their child's emotions. These skills help children to understand and regulate their emotions. As per the Tuning in to Kids manual, two trained, licensed health professionals will co-facilitate each group.
  Arms: Tuning in to Kids (Treatment Arm)

SUMMARY:
The goal of this clinical trial is to learn if a virtually-delivered, group-based psychological intervention, called Tuning in to Kids, is feasible and acceptable for parents of children aged 3 to 6 years with congenital heart disease. The main questions this study aims to answer are:

* What do parents of children with congenital heart disease think of the Tuning in to Kids intervention?
* Is the intervention helpful for parents?
* Is the intervention easy for parents to take part in?
* Do the researchers find it easy or difficult to deliver the Tuning in to Kids intervention to parents of children with congenital heart disease?

Participants will:

* Fill out 3 online surveys at home.
* Take part in the Tuning in to Kids intervention (which includes six 90-minute, weekly, online group sessions and two booster sessions) or standard cardiac care.
* Take part in an interview.

DETAILED DESCRIPTION:
Mental health conditions are common among children with congenital heart disease (CHD) and are strongly associated with cardiovascular morbidity and mortality, as well as lower quality of life. Despite increasing awareness, the mental health needs of children with CHD remain largely unmet, especially among those from historically marginalized and underserved communities. To address this gap, this study will test, for the first time in CHD, a virtually-delivered, group-based psychological intervention, called Tuning in to Kids, designed to teach parents how to help their children understand, regulate, and manage their emotions. The intervention includes six, 90-minute, weekly, online group sessions and two 'booster' sessions, coupled with educational resources and home practice activities to improve parent-child interactions, and enhance child emotional and behavioral functioning. Each group is facilitated by two qualified health professionals who are trained in, and certified to deliver, the Tuning in to Kids intervention. In this pilot randomized controlled trial, we will enroll 40 parents (or other primary caregivers) of children aged 3 or 6 years with CHD who underwent surgical intervention in infancy. The primary aim of this study is to assess intervention acceptability and feasibility, and the results generated will directly inform the design of, and provide preliminary data for, a multicenter efficacy trial to examine short- and longer-term intervention effects.

ELIGIBILITY:
Inclusion Criteria:

1. Child is aged between 3 and 6 years.
2. Child is receiving care from the Cincinnati Children's Heart Institute (at least one cardiology visit in the past 12 months).
3. Child has congenital heart disease requiring cardiopulmonary bypass during infancy (i.e., by age 12 months).
4. Parent or primary caregiver can give consent and participate in the study in English.

Exclusion Criteria:

1. Child has a diagnosed neurodevelopmental disorder (e.g., autism, Trisomy 18), is not speaking, or is not functioning at the developmental level of a typical 3-year-old at the time of study recruitment.
2. Child current medical status or treatment precludes study participation.
3. Parent is aged under 18 years.
4. Parent is currently participating in another parent-focused or parent training program (e.g., Parent-Child Interaction Therapy).
5. Parent suffers from substance misuse or severe, unmanaged mental illness.
6. Parent has an intellectual disability impacting capacity to independently provide informed consent.
7. The child's treating physician or the study interventionalist identifies the parent or child as having a condition or circumstance that is contraindicative to engagement with the Tuning in to Kids program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Enrollment Rate | Enrollment
  ≥70% of eligible approached parents enrolled.
Retention Rate | From enrollment to 1-month post intervention period (up to approximately 12 weeks)
  ≥80% of parents who complete all study procedures.
Proportion of Participants Who Receive All Intervention Content (Fidelity) | From enrollment to 1-month post intervention period (up to approximately 12 weeks)
  ≥80% of parents who receive all intervention content (intervention group only).
Proportion of Participants with Complete Data (Assessment Completion) | From enrollment to 1-month post intervention period (up to approximately 12 weeks)
  ≥80% of parents with complete data.
Intervention Acceptability | After Tuning in to Kids Session 3
  Treatment Acceptability Scale (TAS) score ≥28 (intervention group only). TAS total scores can range from 7 to 56, with higher scores indicating greater intervention acceptability.
Satisfaction with the Intervention | After Tuning in to Kids Session 6 (at approximately 8 weeks)
  Tuning in to Kids Experiences Scale (intervention group only): study-specific measure designed to assess participant satisfaction with the Tuning in to Kids program.

OTHER OUTCOMES:
Child Strengths and Difficulties | From enrollment to 1-month post intervention period (up to approximately 12 weeks)
  Strengths and Difficulties Questionnaire (SDQ): 25-item, validated, widely-used behavioral screening measure with a mix of positive and negatively phrased items assessing five domains (emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, pro-social behavior). Subscale scores are combined (excluding the pro-social scale) into a Total Difficulties score ranging from 0 to 40, with higher scores indicating more problems (with the exception of the pro-social behavior subscale).
Parent Difficulties with Emotion Regulation | From enrollment to 1-month post intervention period (up to approximately 12 weeks)
  Difficulties with Emotion Regulation Scale - Short Form (DERS-SF): 18-item, widely-used, validated scale assessing emotional regulation reported by adults (i.e., parents and caregivers) across 6 domains (strategies, non-acceptance, impulse, goals, awareness, clarity). Response options range from 1 ('almost never') to 5 ('almost always'), with total scores ranging from 18 to 90, and higher scores indicating greater difficulties in emotion regulation.
Parent Emotional Style | From enrollment to 1-month post intervention period (up to approximately 12 weeks)
  Parent Emotional Style Questionnaire (PESQ): Validated 21-item scale assessing parents' beliefs about their child's emotions, including sadness, anger, and fear.
Parent Coping with Children's Negative Emotions | From enrollment to 1-month post intervention period (up to approximately 12 weeks)
  Coping with Children's Negative Emotions Scale (CCNES): 12 scenarios of child negative emotion; parents rate their likelihood of responding in each of six ways.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine A Kasparian, PhD, Principal Investigator — Cincinnati Children's Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data that underlie the results reported in the published paper, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 12 months and ending 24 months following publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
URL: https://www.cincinnatichildrens.org/Kasparian-Lab